CLINICAL TRIAL: NCT06625554
Title: Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection In Assiut University Children Hospital
Brief Title: Urinary Tract Infection In Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed fathy Mohamed farag, Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection In Assiut University Children Hospital, Assiut University
Other Study IDs: UTI in children
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Urinary Tract Infections in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection In Assiut University Children Hospital

DETAILED DESCRIPTION:
Urinary tract infection is the third most common serious bacterial infection in childhood and has been identified as an important risk factor for the development of progressive renal impairment and longterm consequences.

The epidemiology of UTI during childhood varies by age, gender, circumcision status, and other factors. Boys are more susceptible during the first year of life, mostly in the first 3 months, among boys, uncircumcised infants have an eightfold higher risk; due to phimosis, limiteUrinary tract infection is the third most common serious bacterial infection in childhood and has been identified as an important risk factor for the development of progressive renal impairment and longterm consequences.

The epidemiology of UTI during childhood varies by age, gender, circumcision status, and other factors. Boys are more susceptible during the first year of life, mostly in the first 3 months, among boys, uncircumcised infants have an eightfold higher risk; due to phimosis, limited retraction of the foreskin is significantly associated with an increase in UTIs in male infants, afterward, the incidence is mainly higher in girls, due to differences in anatomy .About 5% of girls and 2% of boys experience at least one incident of UTI up to the age of 7 years.

Symptoms of UTI may be minimal and non-specific in infants and small children. Febrile children not suspected of having UTI are as likely to have UTI as those who are suspected of having UTI. Therefore, diagnosis of UTI can not be made on symptomatology alone and urine examination is advocated in children with minimal suspicion of UTI.

Etiological agents of UTI are variable and usually depend on time, geographical location and age of patients. However, Escherichia coli, Proteus mirabilis, Enterobacter agglomerans, Citrobacter frreundii and Klebsiella pneumonia account for over 70% of cases.

According to sex and age, the incidence and clinical symptoms vary, and the causative organisms are different in pediatric UTI. In addition, as antibiotic-resistant pathogens change and are increased due to the abuse of antibiotics and inappropriate selection, it is necessary to select proper antibiotics in the early phase of treatment. Thus, regular antibiotic sensitivity results from the evaluation of UTI are important to improve the effectiveness of treatment.

The gold standard for the diagnosis of UTI is the detection of the pathogen in urine. The pathogen is detected and identified in urine which contributes to antibacterial treatment. Rapid administrations of empirical antibiotics are required before urine culture testing. Meanwhile, complicated UTI often increase the prevalence of inappropriate antibacterial treatment, which in turn increases antibiotic resistance ABR. In pediatric UTI, ABR is also being raised as a clinical challenge. Therefore, there is an urgent need to identify which bacterial strains in children and explore their susceptibility to commonly used antimicrobials. It could guide effective antibacterial therapy and reduce the multi-drug resistance prevalence in children.

In our study we will collect the age, sex, clinical characteristics for children, microorganism isolation and antimicrobial susceptibility profile in children who had been diagnosed with UTI.

According to sex and age, the incidence and clinical symptoms vary, and the causative organisms are different in pediatric UTI. In addition, as antibiotic-resistant pathogens change and are increased due to the abuse of antibiotics and inappropriate selection, it is necessary to select proper antibiotics in the early phase of treatment. Thus, regular antibiotic sensitivity results from the evaluation of UTI are important to improve the effectiveness of treatment.

The gold standard for the diagnosis of UTI is the detection of the pathogen in urine. The pathogen is detected and identified in urine which contributes to antibacterial treatment. Rapid administrations of empirical antibiotics are required before urine culture testing. Meanwhile, complicated UTI often increase the prevalence of inappropriate antibacterial treatment, which in turn increases antibiotic resistance ABR. In pediatric UTI, ABR is also being raised as a clinical challenge. Therefore, there is an urgent need to identify which bacterial strains in children and explore their susceptibility to commonly used antimicrobials. It could guide effective antibacterial therapy and reduce the multi-drug resistance prevalence in children.

In our study we will collect the age, sex, clinical characteristics for children, microorganism isolation and antimicrobial susceptibility profile in children who had been diagnosed with UTI.

ELIGIBILITY:
Inclusion Criteria:

* 1-Children over 1 month and less than 18 year of age. 2-Diagnosed cases of Urinary Tract Infection. 3-who accepted to participate in the study.

Exclusion Criteria:

* 1-neonates and patients more than 18 year. 2-children with chronic kidney diseases. 3-who refused to participate in our study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection In Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sample size | Baseline
  75 patient
  The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is to assess Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection in Children of Assiut University Hospital Based on previous studies (7) the prevalence of antibiotic resistance in children with UTI was 13%, and based on the percentage confidence limits of 5% and a Confidence level=80%
Investigations | Baseline
  1_urine analysis 2- complete blood count(CBC) 3- urine culture and sensitivity
History | Baseline
  1. fever
  2. burning micturation
  3. dysuria
  4. urgency

REFERENCES:
- [Result] Rai GK, Upreti HC, Rai SK, Shah KP, Shrestha RM. Causative agents of urinary tract infections in children and their antibiotic sensitivity pattern: a hospital based study. Nepal Med Coll J. 2008 Jun;10(2):86-90. PMID 18828428
- [Result] Fenta A, Dagnew M, Eshetie S, Belachew T. Bacterial profile, antibiotic susceptibility pattern and associated risk factors of urinary tract infection among clinically suspected children attending at Felege-Hiwot comprehensive and specialized hospital, Northwest Ethiopia. A prospective study. BMC Infect Dis. 2020 Sep 16;20(1):673. doi: 10.1186/s12879-020-05402-y. PMID 32938424
- [Result] Antibiotic Sensitivity Pattern and Demographic Characteristics of Urinary Tract Infection among Hospitalized Children. Saudi J Biomed Res, 7(12): 332-338.